CLINICAL TRIAL: NCT06060496
Title: Theta Burst Stimulation for Alcohol Use Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gopalkumar Rakesh (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Gopalkumar Rakesh, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 86853; 2P30CA177558-11 (NIH)
Record Dates: First submitted 2023-09-22; First posted 2023-09-29 (Actual); Results first posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Alcohol Use Disorder
Keywords: Transcranial magnetic stimulation (TMS)
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Masking Description: Using the MagVenture A/P coil
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Active cTBS and sham cTBS (Experimental): There is only one arm in this study and all participants in this arm will receive 2 interventions: active and sham cTBS in a within subject blinded fashion. They will first receive active cTBS and then sham cTBS, separated by four weeks to minimize carryover effects.
  Interventions: Device: Active cTBS; Device: Sham cTBS

INTERVENTIONS:
Device: Active cTBS — Two cTBS sessions (each session delivering 3600 pulses) separated by 50 minutes
  Other Names: Continuous theta burst stimulation
Device: Sham cTBS — Two sham cTBS sessions (sham mimics the experimental session but does not deliver any electricity to the brain) separated by 50 minutes
  Other Names: Continuous theta burst stimulation

SUMMARY:
The study will examine the effects of two continuous theta burst stimulation (cTBS) sessions (given in a single day) on resting state functional MRI (fMRI), alcohol cue related attentional bias and alcohol craving in patients with alcohol use disorder (AUD).

DETAILED DESCRIPTION:
Although pharmacotherapy and behavioral treatments have been approved for AUD, their effects sizes are modest. Noninvasive neuromodulation like Transcranial magnetic stimulation (TMS) can offer an alternative treatment option for AUD. TMS is a method of noninvasive neuromodulation that utilizes a magnetic field to focal electrical current in the brain. When these electrical currents are focused on specific brain regions, pertinent to the neurobiology of AUD it leads to modulation of behavior and plausibly decrease in alcohol craving and use. Previous TMS studies have used heterogenous parameters, including frequencies ranging from 1 Hz to 20 Hz. Regions targeted by these studies encompassed ventromedial prefrontal cortex, left dorsolateral prefrontal cortex (left dlPFC) and right dorsolateral prefrontal cortex. Two studies used a TMS paradigm with greater efficiency than other routine TMS paradigms, called continuous theta burst stimulation. These studies delivered 3600 pulses of cTBS to the left frontal pole/ventromedial prefrontal cortex and showed significant reduction in alcohol cue reactivity and corroborative changes in both resting state and task based functional connectivity. Of these two studies, one was notable in comparing active cTBS (3600 pulses per session, one session every day for ten days over two weeks) versus sham cTBS. A deep TMS (dTMS) study that compared dTMS (15 sessions, five sessions every week for three weeks) to sham dTMS using an H7 coil (targeting medial prefrontal and anterior cingulate cortices). This study showed decreased craving after treatment and percentage of heavy drinking days in the active versus sham control group. Active dTMS was associated with decreased resting-state functional connectivity of the dorsal anterior cingulate cortex with the caudate nucleus and decreased connectivity of the medial prefrontal cortex to the subgenual anterior cingulate cortex. No study has done multiple sessions of cTBS in a single day. In addition, no study has previously delivered cTBS to the left dlPFC, to modulate alcohol craving and alcohol cue based attentional bias.

ELIGIBILITY:
Inclusion criteria.

* Patients seen at a clinic within the University of Kentucky Healthcare
* 21-60 years of age
* male or female gender
* Able to read, understand and communicate in English
* willing to adhere to the general rules of the UK Healthcare
* Must fulfill criteria for moderate alcohol use disorder.

Exclusion criteria

* Positive pregnancy test for females
* traumatic brain injury, history of seizure disorder, history of or current diagnosis of schizophrenia
* intracranial metal shrapnel
* previous adverse effect with TMS
* sub-threshold consistency while performing behavioral tasks
* failure to show baseline attentional bias to alcohol versus neutral cues.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gopalkumar Rakesh, PhD, Principal Investigator — University of Kentucky
Locations (1):
- 245 Fountain Court, Lexington, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active cTBS and Sham cTBS
Started | 8
Completed | 4
Not Completed | 4
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Active cTBS and Sham cTBS
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 7
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants] — Kentucky, United States
  Participants
    United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Penn Alcohol Craving Scale
Description: Craving measured using the Penn alcohol craving scale (PACS) that has five items and is rated on a scale of 1 to 6. Minimum score is 1 and maximum score is 30. Higher score equates to increased craving
Time Frame: Before and after two cTBS sessions, approximately 2 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- cTBS and Sham cTBS: All participants received both cTBS and sham cTBS in a within subject design
Arm/Group | cTBS and Sham cTBS
Number analyzed (Participants) | 4
units on a scale
  Baseline_cTBS | 11.50 (9.68)
  After second session_cTBS | 11.75 (9.43)
  Baseline_sham cTBS | 8.25 (5.44)
  After second session_sham cTBS | 7.25 (6.70)

2. Primary Outcome: Change in Alcohol Cue Attentional Bias
Description: Fixation time on alcohol cues measured using an eye tracker in milliseconds. Higher score indicates greater attentional bias.
Time Frame: Before and after two cTBS sessions, approximately 2 hours
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- cTBS and Sham cTBS: All participants received cTBS and sham cTBS in a within subject design
Arm/Group | cTBS and Sham cTBS
Number analyzed (Participants) | 4
milliseconds
  Baseline_cTBS | 294.92 (667.18)
  After second session_cTBS | 459.60 (1618.57)
  Baseline_sham cTBS | 355.3 (659.06)
  After second session_sham cTBS | 666.30 (1592.36)

3. Secondary Outcome: Resting State Functional Connectivity
Description: Number of participants with resting state functional connectivity scans acquired before and after cTBS and sham cTBS
Time Frame: Before and after two cTBS sessions, approximately 2 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Active cTBS and Sham cTBS
Number analyzed (Participants) | 4
Participants | 4

ADVERSE EVENTS:
Time Frame: 8 weeks
Groups:
- cTBS and Sham cTBS: All participants received cTBS and sham cTBS in a within-participant design
Arm/Group | cTBS and Sham cTBS
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-03-19): https://cdn.clinicaltrials.gov/large-docs/96/NCT06060496/Prot_SAP_ICF_001.pdf